CLINICAL TRIAL: NCT05361525
Title: Lipoabdominoplasty With Anatomic Definition Versus Traditional Abdominoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Salah El Din Mohamed Hassan, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lipoabdominoplasty
Record Dates: First submitted 2022-04-18; First posted 2022-05-04 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Abdomen Enlarged

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipoabdominoplasty with anatomic definition (Active Comparator): Lipoabdominoplasty with anatomic definition without over dissection on the lateral recti region
  Interventions: Procedure: modified saldhana's technique
- traditional abdominoplasty (Sham Comparator): abdominoplasty with dissection in v- shaped pattern till coastal margin
  Interventions: Procedure: Traditional abdominoplasty

INTERVENTIONS:
Procedure: modified saldhana's technique — tummy tuck with anatomic definition using liposuction
  Arms: Lipoabdominoplasty with anatomic definition
Procedure: Traditional abdominoplasty — uses the traditional technique of abdominoplasty with liposuction with v-shaped dissection till the coastal margin
  Arms: traditional abdominoplasty

SUMMARY:
A tummy tuck also known as abdominoplasty is a cosmetic surgical procedure to improve the shape and appearance of the abdomen.

DETAILED DESCRIPTION:
Lipoabdominoplasty guarantees a safe combination of abdominoplasty and liposuction while minimizing the risk of ischemic flap complications. This is because of the limited undermining performed and the liposuction adjunct, both of which minimize perforator injury. In the last several years, the integration of anatomic definition through the use of liposuction has further refined the procedure, led to improved results, and increased patient satisfaction. The more natural results of the anatomic abdominal definition is a next step in abdominal contour refinement.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 25 to 60 with redundant abdominal wall.
* BMI less than 35.

Exclusion Criteria:

* Patients younger than 25 or older than 60.
* BMI more than 35.
* Hernias and scars interfering with abdominal vascularity.
* Patients smoking or with comorbidities (DM, HTN, ...etc).
* Patients seeking for another pregnancies.
* Any causes that may interfere with general anaesthesia. Refusal for any part of the written conset

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Aesthetically | 6 months post op
  natural look, patient satisfaction on scale (Rosenberg self esteem scale, it uses scale 0-30, where score less than 15 indicate low self esteem problem) with 10 items 6 months post operative and compare it with the preoperative results of the same patient, patient sexual satisfaction after 6 months in comparison with the preoperative results, doctors opinion and natural curves at the muscle insertion sites

SECONDARY OUTCOMES:
complications | up to 2 weeks post operatively
  the usual complications of abdominoplasty

CONTACTS AND LOCATIONS:
Locations (1):
- Asyut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Lipoadominoplasty with anatomin definition versus traditional abdominoplasty
Supporting Information: Study Protocol, SAP, ICF
Time Frame: it will be available after the study is complete in approximately two years
Access Criteria: access for every one